CLINICAL TRIAL: NCT05315661
Title: Clinical Assessment on the Safety and Potential Efficacy of Mesenchymal Stem Cells Preconditioned With Ethionamide (ET-STEM) in Patients With Frontotemporal Dementia (FTD)
Brief Title: The Safety and The Efficacy Evaluation of ET-STEM in Patients With Frontotemporal Dementia
Acronym: FTD_ET-STEM
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Hee Jin Kim, assistant professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-02-089
Record Dates: First submitted 2022-03-01; First posted 2022-04-07 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Frontotemporal Dementia
MeSH Terms: conditions — Frontotemporal Dementia

STUDY DESIGN:
Intervention Model Description: Single Group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): injected with 3x10^7 cells/2mL of ET-STEM to intraventricular space via an Ommaya reservoir. repeated 3 times at 4 week intervals
  Interventions: Drug: ET-STEM

INTERVENTIONS:
Drug: ET-STEM — mesenchymal stem cells preconditioned with ethionamide

SUMMARY:
The primary purpose of this study is to evaluate the safety and the tolerability of 3 repeated doses of ET-STEM (Mesenchymal stem cells preconditioned with ethionamide) in patients with FTD.

DETAILED DESCRIPTION:
Subjects with FTD, who signed the informed consent form and meet the eligibility criteria will undergo Ommaya reservoir insertion. 2 weeks after Ommaya reservoir insertion, the subjects will be injected with 3x10^7 cells/2mL of ET-STEM to intraventricular space via an Ommaya reservoir. The injection will be repeated 3 times at 4 week intervals. The subjects will be hospitalized for 24 hours and observed for acute adverse events. 4 weeks after the 3rd injection, safety and potential efficacy will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Korean male or female at 40-85 years of age
2. Diagnosis of one of the 3 subtyes of FTD according to the diagnostic criteria for 3 subtypes of FTD

   ① Probable bvFTD (behavior variant FTD)

   ② svPPA (semantic variant primary progressive aphasia)

   ③ nfvPPA (nonfluent/agrammatic variant primary progressive aphasia)
3. K-MMSE ≥ 10
4. Subjects with trusted caregivers who regularly contact the subjects and can accompany the subjects when visiting the hospital.
5. Negative result of amyloid PET imaging
6. A subject who is informed of the clinical trial and signs a consent form (If unable to sign, a consent from a legally acceptable representative is required)

Exclusion Criteria:

1. Subjects with dementia cause by other than FTD (i.e. infection of central nervous system, Creutzfeld-Jacob disease, severer head trauma, Huntington's disease, Parkinson's disease, Alzheimer's disease and vascular dementia)
2. Subjects with psychological disorder. (i.e. depression, schizophrenia , bipolar disorder, etc) (except for subjects who were misdiagnosed with psychological disease due to the initial neuropsychiatric symptoms of FTD)
3. Subjects with uncontrolled hypotension, hypertension, diabetes and thyroid disease.
4. Subjects with a cancer (including brain tumor)
5. Subjects with bleeding disorder
6. Woman of childbearing age who refused to practice medically acceptable contraceptive method (post menopausal patient with no menstruation for at least 12 months is considered as infertile)
7. Pregnant or lactating females
8. History of stroke within 3 months prior to study enrollment
9. Substance/alcohol abuse 1
10. Contraindicated for any of the tests performed during the clinical trial period(for example, MRI, CT,PET)
11. A subject in whom Ommaya reservoir insertion and general anesthesia are considered difficult
12. Abnormal Laboratory findings at Screening
13. Suspected active lung disease based on chest X-ray at Screening
14. Positive hepatitis B nuclear antibody and hpatitis C antibody
15. Subjects who the principal investigator considers inappropriate for participation in the study due to the possible harmful effect on the subjects,difficulty in study completion, or previous or current medical conditions that may disturb evaluation of study results
16. Subjects who the principal investigator considers impossible to comply with clinical research procedures.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-07-06 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
To determine DLT (Dose limiting toxicity) | First 3-week cycle of treatment
  incidence rate of DLT (Dose limiting toxicity)
adverse events as assessed by CTCAE v5.0 | up to 5years
  all potentially treated subjects to assess the safety

SECONDARY OUTCOMES:
ADAS-Cog 13 response rate | Screening, after the first administration12weeks, 48weeks, 96weeks, 144weeks, 192weeks, 240weeks
  response rate, no change or improvement on ADAS cog 13 score
The Clinical Dementia Rating Sum of Boxes | Screening, after the first administration12weeks, 48weeks, 96weeks, 144weeks, 192weeks, 240weeks
  Change from the baseline in CDR-SB, min 0, max 24, higher scores mean a worse outcome
Alzheimer's Disease Cooperative Study- instrumental items of the Activities of Daily Living Inventory | the first administration12weeks, 48weeks, 96weeks, 144weeks, 192weeks, 240weeks
  Change from the baseline in ADCS-iADL, min 0, max78, higher scores mean a better outcome
Caregiver-administered Neuropsychiatric Inventory | the first administration12weeks, 48weeks, 96weeks, 144weeks, 192weeks, 240weeks
  Change from the baseline in CGA-NPI, min 0, max 144, higher scores mean a worse outcome
preliminary efficacy | up to 12weeks
  Change from the baseline in CSF biomarkers
K-MMSE | the first administration12weeks, 48weeks, 96weeks, 144weeks, 192weeks, 240weeks
  Korean Mini-Mental State Examination(MMSE), min 0, max 30, higher scores mean a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: HeeJin Kim, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, Gangnam-gu, South Korea

IPD SHARING:
Plan to Share IPD: No